CLINICAL TRIAL: NCT04115670
Title: Influence of Health Determinants and Therapeutic Alliance on the Effectiveness of a Pain Neuroscience Education Combined With Motor Control Training With Neurocognitive Focus on Chronic Lumbar Pain in a Population of Professional Caregivers
Brief Title: Influence of Health Determinants on Physical Exercise Therapy With a Neurocognitive Focus on Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundació Universitària del Bages (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UManresa_Caregivers2019
Record Dates: First submitted 2019-10-01; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Chronic Low-back Pain
MeSH Terms: interventions — Exercise; Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- specific intervention (experimental) (Experimental): Specific intervention (experimental). The intervention group will carry out 3 sessions of specific pain education + 15 sessions of physical training.
  Interventions: Behavioral: Group of educational intervention on the neurophysiology of pain and physical exercises
- control group (no intervention) (Active Comparator): NO intervention
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Group of educational intervention on the neurophysiology of pain and physical exercises — The physiotherapist of the institution will execute the intervention on the group:
  * 3 first pedagogical sessions on the neurophysiology of pain, distributed: 1 group session, 1 individual session at home, 1 in a personal interview format. These 3 sessions will last 2 weeks to be completed.
  * Afterward, the protocol of physical exercise training will begin, supervised by the same physiotherapist who carried out the three initial sessions. There will be 15 sessions of specific and individualized physical exercise, in small groups of maximum 5 people. The duration of this part will be 10 weeks, so that from week 1 to 5 is 2 times per week, and from week 6 to 10 just 1 time per week.
  Arms: specific intervention (experimental)
Behavioral: Control group — The control group will follow its normal course of activity
  Arms: control group (no intervention)

SUMMARY:
Protocols in which pain neuroscience education is combined with physical exercise have shown recently greater effectiveness in the treatment of low back pain in comparison to protocols based only on one of the two approaches. The professional caregiver has a high incidence of low back pain related to the specific aspects of this collection with the low physical condition, the typical tasks performed and other psychosocial aspects. Individual characteristics of these caregivers may condition the effectiveness of the therapy as well as demographic aspects or the alliance between patient and physiotherapist. The aim of this study is to determine the influence of certain health determinants on the effectiveness of a therapy that combines pain neuroscience education and motor control training from a neurocognitive perspective on chronic low back pain in a population of professional caregivers in Bages, analyzing the reduction of low back pain, the improvement of functionality, the reduction of muscle movement and the improvement of muscle coordination.

It will be a quasi-experimental pre-post design, prospective, with a control group, lasting 3 months. The intervention will be performed using a sample of professional caregivers, and the data will be collected before the intervention, at the end of the intervention, and 3-6 months after the intervention. Pain, functionality, conducts of fear/avoidance, and muscular coordination will be analyzed

ELIGIBILITY:
Inclusion Criteria:

* Of legal age
* Participants who present lumbar or lumbosacral pain all the time for more than 1 year
* Score of 6 on the Visual Analogical Scale
* Have been at work (same position) longer than 1 year

Exclusion Criteria:

* Other alterations and diseases of the musculoskeletal system that may interfere with the results of the intervention.
* Pregnancy during the study time
* Older than 65 years old

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12-02 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-12-20 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Pain perceived at 3 months: Visual Analogue Scale | Baseline and 3 months
  Analisis of pain, using the Visual Analogue Scale, that measure from 0 (no pain) to 10 (excruciating pain)
Change from Baseline in Pain perceived at 6 months: Visual Analogue Scale | Baseline and 6 months
  Analisis of pain, using the Visual Analogue Scale, that measure from 0 (no pain) to 10 (excruciating pain)

SECONDARY OUTCOMES:
Change from Baseline in Fear and avoidance of movement at 3 months | Baseline and 3 months
  Tampa Scale of Kinesophobia, a scale with 11 items, the rating ranges from 11 points to 44 points. A high value indicates that there is a high degree of fear of movement.
Change from Baseline in Pain disability at 3 months: Oswestry Disability Index | Baseline and 3 months
  Oswestry Disability Index, This scale consists of 10 questions, each of them with answers graduated from 0 (no relevant) to 5 (very relevant), from which the % of disability of the individual is obtained from the formula: Total points of the answers / 50 *100= % disabled

CONTACTS AND LOCATIONS:
Overall Officials: Júlia Jubany, PhD, Principal Investigator — University of Vic - Central University of Catalonia
Locations (1):
- Universitat de Vic-Universitat de Catalunya (UVic-UCC), Manresa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data about the protocol intervention, primary outcome measures and final report will be available for the Institution director.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Before the intervention starts
Access Criteria: Only for institution director

REFERENCES:
- [Background] Hoy D, Bain C, Williams G, March L, Brooks P, Blyth F, Woolf A, Vos T, Buchbinder R. A systematic review of the global prevalence of low back pain. Arthritis Rheum. 2012 Jun;64(6):2028-37. doi: 10.1002/art.34347. Epub 2012 Jan 9. PMID 22231424
- [Background] Radebold A, Cholewicki J, Panjabi MM, Patel TC. Muscle response pattern to sudden trunk loading in healthy individuals and in patients with chronic low back pain. Spine (Phila Pa 1976). 2000 Apr 15;25(8):947-54. doi: 10.1097/00007632-200004150-00009. PMID 10767807
- [Background] Kamper SJ, Apeldoorn AT, Chiarotto A, Smeets RJ, Ostelo RW, Guzman J, van Tulder MW. Multidisciplinary biopsychosocial rehabilitation for chronic low back pain. Cochrane Database Syst Rev. 2014 Sep 2;2014(9):CD000963. doi: 10.1002/14651858.CD000963.pub3. PMID 25180773
- [Background] Malfliet A, Kregel J, Meeus M, Cagnie B, Roussel N, Dolphens M, Danneels L, Nijs J. Applying contemporary neuroscience in exercise interventions for chronic spinal pain: treatment protocol. Braz J Phys Ther. 2017 Sep-Oct;21(5):378-387. doi: 10.1016/j.bjpt.2017.06.019. Epub 2017 Jul 8. PMID 28736211
- [Background] Yang H, Haldeman S, Lu ML, Baker D. Low Back Pain Prevalence and Related Workplace Psychosocial Risk Factors: A Study Using Data From the 2010 National Health Interview Survey. J Manipulative Physiol Ther. 2016 Sep;39(7):459-472. doi: 10.1016/j.jmpt.2016.07.004. Epub 2016 Aug 25. PMID 27568831